CLINICAL TRIAL: NCT02761356
Title: The Added Value of Hybrid Functional Anatomical Imaging PET-CT and SPECT-CT in Patients Treated With Yttrium-90 SIRT for Liver
Brief Title: The Added Value of Hybrid Functional Anatomical Imaging PET-CT and SPECT-CT in Patients Treated With Y-90 SIRT for Liver Malignancies
Status: Completed | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: TASMC-16-ES-0413-15-TLV-CTIL
Record Dates: First submitted 2016-02-11; First posted 2016-05-04 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Primary Liver Tumor, Metastatic Liver
MeSH Terms: interventions — technetium Tc 99m-Sn aggregated albumin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Tc99-MAA and SPECT-CT: 26 of the patients were examined with Tc99-MAA and SPECT-C
  Interventions: Other: Tc99-MAA
- Tc99-MAA , SPECT-CT and PET-CT: 24 patients were examined with Tc99-MAA , SPECT-CT and PET-CT.
  Interventions: Other: Tc99-MAA

INTERVENTIONS:
Other: Tc99-MAA — To evaluate the fisibility of Tc99-MAA injected intra epatic artery to predict uptake of Yttrium-90 SIRT in patients with liver malignancies
  Other Names: Tc-99m-macroaggregated albumin

SUMMARY:
Patients cohort is composed of 50 consecutive patients both male and female with hepatic malignancies, refered to our nuclear medicine department in the process of radioembolization between January 2010- August 2015. 26 of the patients were examined with Tc99-MAA and SPECT-CT and 24 patients were examined with Tc99-MAA , SPECT-CT and PET-CT. Our study protocol was as follows:

1. Collection of anamnestic data
2. Calculation of liver tumor volume with quantification software
3. Evaluation of the liver tumor involvement
4. Evaluation of liver to lung shunt
5. Calculation dose of SIRTEX
6. Y90 imaging
7. Follow Up

DETAILED DESCRIPTION:
The description of the various stages that the patient goes through SIRTex treatment in the department of nuclear medicine and their roll in the study is as following:

The first stage is dedicated to the evaluation of the patient's illegibility for the treatment.

1. In Angiography department
2. In Nuclear medicine department assessment of liver-lung shunting (planar images). Followed by SPECT-CT of the upper abdomen. SPECT with Low dose CT is used to identify a leak to the stomach, duodenum and mesentery, as well as to assess uptake of Tc-99m-MAA in tumor lesions. In order to increase SPECT-CT resolution and sensitivity we co-registrated SPECT-CT with diagnostic CT provided from previous contrast enhanced CT or PET-CT. In this procedure, the Low dose CT is used as bridge between diagnostic CT and the functional imaging SPECT.
3. Calculation dose of Sirtex therapy. At this stage the purpose of the study will be to investigate the added value of SPECT-CT in the estimation of Tc-99m-MAA uptake in tumor lesions.

The second stage is dedicated to the assessment Y-90-SIRTex uptake in liver tumors and to exclude extra hepatic leak. Several hours after treatment patients perform SPECT-CT using Brummshtrullung emission or PET-CT with the peak Zr-90.

At this stage , in our study, we will compare liver lesions uptake of Tc-99m-MAA in the SPECT-CT to lesions uptake of Y-90 -SIRT SPECT/PET-CT as well as to assess if SPECT-CT withTc-99m-MAA may be used as a predictor of Y-90-SIRTex uptake in liver lesion. Does SPECT-CT with Tc-99m-MAA change patient managment.

The third stage of the study is the collection and monitoring of post treatment outcome data.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18. 2. Patients with malignancy of the liver (metastasis or primary tumor) who were treated with Y90 SIRT and were refered to the nuclear medicine department for a PET-CT.

Exclusion Criteria:

* 1. Age < 18. 2. Pregnant woman 3. Children and legally incompetent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients treated with Yttrium-90 SIRT for liver malignancies
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Visual assesment of Tc-99m-MAA in liver lesions compared to visual assesment of Y-90 sirtex. | one year
  Undestanding the role of Tc-99- MAA in the prediction of Y90 sirt uptake in liver lesions by visual assesment with PET-CT and SPECT-CT imaging

CONTACTS AND LOCATIONS:
Overall Officials: Einat Even-Sapir, Phd, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Department of Nuclear Medicine, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No